CLINICAL TRIAL: NCT06837259
Title: A Phase 1, Open-Label, Fixed-Sequence Study to Evaluate the Effect of OATP Inhibition on the Single Dose Pharmacokinetics of PF-07328948 in Healthy Adult Participants.
Brief Title: A Study to Learn if Study Medicines Called Cyclosporine and Clarithromycin Affect How the Body Processes the Other Study Medicine Called PF-07328948 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: C4921008; 2024-520126-11-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Cyclosporine; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Period 1 (Experimental): PF-07328948
  Interventions: Drug: PF-07328948
- Period 2 (Experimental): cyclosporine and PF-07328948
  Interventions: Drug: PF-07328948; Drug: cyclosporine
- Period 3 (optional) (Experimental): clarithromycin and PF-07328948
  Interventions: Drug: PF-07328948; Drug: clarithromycin

INTERVENTIONS:
Drug: PF-07328948 — single oral dose day 1 and day 12 (Part A) and day 4 (part B)
Drug: cyclosporine — 600 mg capsule day 12 (Part A)
  Arms: Period 2
Drug: clarithromycin — 500 mg tablets twice daily day 1 to day 6 (Part B)
  Arms: Period 3 (optional)

SUMMARY:
The purpose of this study is to learn about the effect of cyclosporine, an immunosuppressant (medicine that suppresses the immune system), on the pharmacokinetics (PK) of PF-07328948 in healthy participants (Part A). The study may also estimate the effect of clarithromycin, an antibiotic, on the PK of PF-07328948 in healthy participants (Part B is optional).

This study is seeking participants who:

* are 18 years of age or older
* are male or female who are not of childbearing potential
* are healthy (do not have a disease) The study will consist of two parts - Part A and Part B.

Part A will consist of two treatments:

* one dose of PF-07328948 solution to be taken by mouth on day 1.
* one cyclosporine 600 mg capsule taken together with a dose of PF-07328948 solution by mouth on day 12.

Before study Part A starts, all participants will go through a screening process which may last for a period of up to 28 days. During this period, the participant's medical history and past and current medications will be reviewed. A series of tests will also be performed.

If the participants meet all required criteria and want to continue, they will be brought into the study clinic to stay overnight for 17 days. During this period, the experiences of participants receiving the study medicine will be examined. Samples for laboratory assessments will be collected. Vital signs and medical assessments will also be performed. This will help determine if it is safe to take the study medicines together and what happens to these medicines in one's body (called PK assessment). After Part A, participants will be discharged from the clinic.

Based upon the results of Part A, study participants may proceed to Part B. If Part B occurs, participants will return to the study clinic and remain in the clinic for 8 days. There will be a gap of at least 7 days between Part A and Part B.

Part B will consist of a third treatment:

- clarithromycin 500 mg tablet to be taken 2 times a day for 6 days. On day 4, the tablet will be taken together by mouth with a dose of PF-07328948 solution.

During this period, similar laboratory and medical assessments as done in Part A will occur. After Part B, participants will be discharged from the clinic.

The participant will be contacted for a follow up visit by telephone about 30 days after final treatment. This is to check up on how the participant is doing and to conclude the study. If only Part A occurs, a participant will be in the study about 44 days. If Part B occurs, a participant will be in the study for about 64 days.

ELIGIBILITY:
Inclusion:

* Males and females (of non-childbearing potential) who are overtly healthy.
* Body mass index of 18.5-35 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm/Hg for participants ≥60 years old, following at least 5 minutes of supine rest. If systolic BP is ≥ 140 or 150 mm Hg (based on age) or diastolic ≥90 mm Hg, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* Evidence of a prothrombotic state (history of deep vein thrombosis, pulmonary embolism, or arterial thrombosis or a known genetic predisposition [Factor V Leiden, prothrombin G20210A, Protein C/S deficiency, antithrombin deficiency])
* An eGFR <60 units mL/min/1.73m², as determined by the CKD-EPI equation using serum creatinine
* Standard 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete left bundle branch block (LBBB), signs of an acute or indeterminate age myocardial infarction, ST segment and/or T wave changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias).
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary: ALT, AST, Bilirubin ≥1.5 x ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of PF-07328948 | Hour 0, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 post-dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of PF-07328948 | Hour 0, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 post-dose
  if data permits
Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUClast) of PF-07328948 | Hour 0, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 post-dose
  If AUCinf cannot be completed

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline (Day 0) up to 35 days after last dose of study medication
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | Baseline up to Day 18 (Part A) or up to Day 35 (optional Part B)
Number of Participants With Clinically Significant Change From Baseline in Blood Pressure and Pulse Rate | Baseline up to Day 18 (Part A) or up to Day 35 (optional Part B)
Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Findings | Baseline up to Day 18 (Part A) or up to Day 35 (optional Part B)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4921008